CLINICAL TRIAL: NCT06460181
Title: Impact of Astaxanthin on Cognition in Recreationally Active Females
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-021
Record Dates: First submitted 2024-05-28; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Mental Fatigue
MeSH Terms: conditions — Mental Fatigue | interventions — astaxanthine

STUDY DESIGN:
Intervention Model Description: Groups will be randomized and parallel. They will not cross-over with each other.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will supplement with either AX or a matched placebo. The dosage of AX (12 mg/day) is FDA approved and will be administered orally by one soft gel capsule. The treatments will be blinded to the participants and the investigator. Treatments will be sorted be an independent party not associated with data collection or analysis.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Astaxanthin (Active Comparator): Astaxanthin will be administered in a dosage of 12 mg/day orally by one soft gel capsule per day. the capsule consist of natural Astaxanthin and olive oil.
  Interventions: Dietary Supplement: Astaxanthin
- Placebo (Placebo Comparator): The placebo will be administered orally by one soft gel capsule per day. The placebo contains olive oil and is color, order, and taste matched to the Astaxanthin soft gels.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Astaxanthin — Manufactured by AstaReal Inc
  Arms: Astaxanthin
Dietary Supplement: Placebo — Manufactured by AstaReal Inc
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the protentional that the antioxidant Astaxanthin has on mitigating cognitive decline following mental fatigue.

DETAILED DESCRIPTION:
Dietary supplements are used in all levels of sports to impact various areas of athletic performance. Prolonged physical activity or cognitive engagement, which is a part of the competition, can increase mental fatigue (MF) such that the athlete begins to experience impaired decision-making skills and slower reaction times, resulting in a less-than-optimal athlete by the end of the competition. Thus, identifying interventions that may preserve an individual's ability to perform following a state of MF would interest individuals often engaged in competition or training.

Astaxanthin (AX) is a naturally occurring antioxidant typically found in marine species such as algae, salmon, trout, and shellfish. AX's unique structure may mitigate inflammation. Cognitively, AX can cross the blood-brain barrier to help support the mitochondria when metabolic or cognitive demands are increased. While there have been promising results in elderly individuals of AX's ability to mitigate reductions in cognitive performance when fatigued. However, investigations in younger, more active individuals are warranted. Therefore, the purpose of this study to examine the impact of four weeks of AX supplementation at 12 mg/day on various markers of cognitive performance following a mental fatiguing protocol in recreationally active females.

The cognitive methods are adapted from another previous study titled, "No Benefit of Ingesting a Low-Dose Ketone Monoester Supplement on Markers of Cognitive Performance in Females" (IRB#: 2023-009). This study is a double-blind between design. Supplementation will last four weeks with each subject will consume either 12 mg/day of AX or a matched placebo. The participants will report to the lab for four separate trials. There will be two cognitive trials before and after supplementation. A 4 week supplementation period will occur after trials 1 & 2, followed by a repeat of these sessions for post-testing. We hypothesize that AX will mitigate cognitive detriments following mental fatigue. The significance of these results may extend to female athletes looking to enhance performance by protecting cognitive ability from declining after fatigue.

Cognitive Protocol: Participants will use software called SOMA NPT to complete a series of validated cognitive tasks that test different aspects of cognition. The cognitive battery of test that will be used includes a Psychomotor Vigilance Test (PVT; 5 min), Task Switching (3 min), and Incongruent Flaker (3 min). The task that will be used to induce mental fatigue is a Time-Loaded-Dual-Back task (TLDB; 15 min). A control video titled World Class Trains (15 min) has been validated to produce no emotional response. Each subject will complete a trial with the mental fatigue protocol and a control before supplementation.

Lipid Panel: A lipid panel to asses participants cholesterol and glucose levels will be taken both pre and post supplementation by using a capillary finger prick.

ELIGIBILITY:
Inclusion Criteria:

* The participant population will be healthy, recreationally active females between the ages of 18-39 without any medical conditions. To be deemed recreationally active, they must meet the World Health Organization minimum activity guidelines of completing at least 150 to 300 min moderate-intensity activity or 75-150 min of vigorous-intensity activity a week, plus muscle-strengthening activities 2 or more days a week.
* Adult females with a stable body weight (± 5 lbs.) for 2 months
* Adult females with a normal menstrual cycle
* Adult females not on a low-carb, high-fat diet or intermittent fasting
* Adult females who are not pregnant of actively attempting to become pregnant

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Reaction time | Pre supplementation and post 4-week supplementation period.
  How quickly the participant reacts to a stimulus. Expressed in millaseconds.
Speed | Pre supplementation and post 4-week supplementation period.
  Speed at which responses are given.
Responses Correct per Second | Pre supplementation and post 4-week supplementation period.
  Accuracy of responses over time.
Mental Fatigue | Pre supplementation and post 4-week supplementation period.
  Assessed using a 180mm visual analog scale. 0mm = no mental fatigue, 180mm = highest possible mental fatigue.

SECONDARY OUTCOMES:
Lipid Panel | Pre and post
  Cholesterol, lipid, and glucose levels. Tested using blood from the capillaries of the fingers

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Alabama, Florence, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT06460181/ICF_000.pdf